CLINICAL TRIAL: NCT02507752
Title: An Observational, Prospective, Multicenter, Local, to Assess the Quality of Life Through the Use of Questionnaires in a Cohort of Patients With Rheumatoid Arthritis Treated With Anti-CD20 Therapy
Brief Title: An Observational Quality of Life Study in Participants With Rheumatoid Arthritis Treated With Rituximab
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22064
Record Dates: First submitted 2015-07-23; First posted 2015-07-24 (Estimated); Results first posted 2015-12-29 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Rituximab: Participants who are receiving 1000 milligrams (mg) intravenous (IV) infusion of rituximab on Day 1 and Day 15 as part of standard of care of the treating site will be included in this observational study.

SUMMARY:
This multicenter prospective observational study will evaluate the quality of life in participants with rheumatoid arthritis (RA) who are initiated with rituximab (MabThera/Rituxan). Participants will be followed for 6 months from initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants of both genders who are 18 years or older
* Diagnosis of RA for at least 6 months according to the criteria of the American College of Rheumatology (ACR) of 1987 for the RA classification
* Participants with medically prescribed or being administered with unique rituximab infusion in the least 3 days, according to the approved label
* Ability to meet the program's requirements and to voluntarily sign the Informed Consent Term.

Exclusion Criteria:

* Participants who have received any investigational medication within less than or equal to (<=) 1 year before the first dose of the currently indicated treatment
* Participants with an active infection
* Participants with conditions that may interfere in the ability to understand the requests of data collection and to obey to the study's requirements
* Functional Class IV defined based on the ACR functionality criteria for RA
* Participants who can not or who do not want, for any reason, to answer the questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with RA initiating rituximab
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2009-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (13):
- Brazil (13):
  - Salvador, Estado de Bahia
  - Cuiaba, Mato Grosso do Sul
  - Juiz de Fora, Minas Gerais
  - Uberlândia, Minas Gerais
  - Curtiba, Paraná
  - Recife, Pernambuco
  - Rio de Janeiro, Rio de Janeiro
  - Porto Alegre, Rio Grande do Sul
  - Campinas, São Paulo
  - Osasco, São Paulo
  - Santo André, São Paulo
  - São José do Rio Preto, São Paulo
  - São Paulo, São Paulo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 95 participants were screened for eligibility between July 2009 and December 2011 at 16 centers in Brazil.
Pre-assignment Details: Out of 95 participants, 72 who answered at least one short form 36 (SF-36) questionnaire made up the Intent-to-treat (ITT) population
Groups:
- Rituximab: Participants with rheumatoid arthritis, who were treated with rituximab according to standard medical practice, were included in this cohort.
Period: Overall Study
Arm/Group | Rituximab
Started | 72
Completed | 55
Not Completed | 17
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 6
Not completed — Lost to Follow-up | 7
Not completed — Infusion reaction at first infusion | 1
Not completed — Participant didn't perform visit Week 12 | 1
Not completed — Participant didn't perform visit Week 24 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are summarized for the ITT population that included all screened participants who answered at least one short form 36 (SF-36) questionnaire.
Arm/Group | Rituximab
Number analyzed (Participants) | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving an Improvement of at Least 0.22 Units in Health Assessment Questionnaire (HAQ) at Week 24
Description: The Health Assessment Questionnaire-Disability Index (HAQ-DI) is a 20-question instrument that assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping and activities of daily living). Responses in each functional area are scored from 0 to 3 (0=no difficulty and 3=inability to perform a task in that area). HAQ-DI total scores expressed as overall mean score with range 0-3: 0-0.25=normal functioning; 0.25-0.5=mild functional limitation; 0.5-1=moderate functional limitation; more than 1=significant functional limitation. The proportion of participants achieving a clinically important reduction of >= 0.22 point in HAQ (disease-specific questionnaire) at Week 24 was evaluated. HAQ was assessed using the set of observed cases (OC) at each assessment time. An improvement of 0.22 units in HAQ-DI was considered to be a clinically significant improvement.
Time Frame: Week 24
Population: The ITT population included all screened participants who answered at least one SF-36 questionnaire.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Rituximab
Number analyzed (Participants) | 38
Percentage | 57.9 [42.2 to 72.1]

2. Primary Outcome: Mean Change From Baseline in the Short-Form (SF-36) Health Survey Physical Component Score and Mental Component Score at Week 24
Description: SF- 36 investigates the standard of quality of life through a general health assessment and not specific to a particular disease, age or treatment group. It is a 36-item questionnaire measuring 8 domains (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health). Each domain score ranges from 0 (worst) to 100 (best), with higher scores reflecting better health-related functional status. Two summary scale scores were computed based on weighted combinations of the 8 domain scores: the Physical Component Summary and the Mental Component Summary. SF-36 was assessed using the set of observed cases (OC) at each assessment time.
Time Frame: Baseline and Week 24
Population: The ITT population included all screened participants who answered at least one SF-36 questionnaire. n = number of participants analyzed for a given component of SF-36.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Rituximab
Number analyzed (Participants) | 72
scores on a scale
  Physical component score, n = 36 | 14.6 (2.5)
  Mental component score, n = 38 | 9.8 (3.8)
Statistical Analysis 1: Comparison: Rituximab; Physical component score at Week 24: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Rituximab; Mental component score at Week 24: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p = 0.014, ANOVA

3. Secondary Outcome: Number of Participants With Infusion Reactions, Infectious Events and / or Other Adverse Events in the 24 Weeks After the Start of Treatment.
Description: An infusion reaction is defined as an adverse event that occurs during infusion or within 24 hours after infusion of Rituximab. All infectious events, whether considered related or not to Rituximab, were collected for the safety analysis of the study. An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Time Frame: Up to 24 Weeks
Population: The ITT population included all screened participants who answered at least one SF-36 questionnaire.
Measure: Number; unit: participants
Arm/Group | Rituximab
Number analyzed (Participants) | 72
participants
  Infusion reactions | 15
  Infectious events | 5
  Adverse events | 21

4. Secondary Outcome: Mean Change From Baseline in Erythrocyte Sedimentation Rate (ESR)
Description: Erythrocyte Sedimentation Rate is an acute phase reactant and a measure of inflammation.
Time Frame: Baseline, Week 12, Week 24
Population: The ITT population included all screened participants who answered at least one SF-36 questionnaire. n = the number of participants analyzed at the given time point.
Measure: Mean (Standard Error); unit: mm/hr
Arm/Group | Rituximab
Number analyzed (Participants) | 72
mm/hr
  Week 12 (n = 48) | -7.5 (3.1)
  Week 24 (n = 46) | -11.5 (3.7)
Statistical Analysis 1: Comparison: Rituximab; Mean change from Baseline in ESR at Week 12: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p = 0.021, ANOVA
Statistical Analysis 2: Comparison: Rituximab; Mean change from Baseline in ESR at Week 24: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p = 0.003, ANOVA

5. Secondary Outcome: Mean Change From Baseline in C-reactive Protein (CRP).
Description: CRP is an inflammation marker. High levels of this protein indicate inflammation in diseases such as Rheumatoid Arthritis.
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 4
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | Rituximab
Number analyzed (Participants) | 72
mg/L
  Week 12 (n = 37) | -0.3 (0.9)
  Week 24 (n = 36) | -0.5 (1)
Statistical Analysis 1: Comparison: Rituximab; Mean change from Baseline in CRP at Week 12: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p = 0.744, ANOVA
Statistical Analysis 2: Comparison: Rituximab; Mean change from Baseline in CRP at Week 24: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p = 0.646, ANOVA

6. Secondary Outcome: Mean Change From Baseline in Swollen Joint Count (SJC)
Description: A swollen joint count is the most specific clinical method to quantify abnormalities in participants with rheumatoid arthritis (RA). It reflects the amount of inflamed synovial tissue.
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Number of swollen joints
Arm/Group | Rituximab
Number analyzed (Participants) | 72
Number of swollen joints
  Week 12 (n = 58) | -5.2 (0.6)
  Week 24 (n = 56) | -5.1 (0.7)
Statistical Analysis 1: Comparison: Rituximab; Mean change from Baseline in SJC at Week 12: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Rituximab; Mean change from Baseline in SJC at Week 24: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p < 0.001, ANOVA

7. Secondary Outcome: Mean Change From Baseline in Tender Joint Count (TJC)
Description: A tender joint count is the most specific clinical method to quantify abnormalities in participants with rheumatoid arthritis (RA). It is associated more with the level of pain.
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Number of tender joints
Arm/Group | Rituximab
Number analyzed (Participants) | 72
Number of tender joints
  Week 12 (n = 58) | -6 (0.8)
  Week 24 (n = 56) | -7 (0.9)
Statistical Analysis 1: Comparison: Rituximab; Mean change from Baseline in TJC at Week 12: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Rituximab; Mean change from Baseline in TJC at Week 24: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p < 0.001, ANOVA

8. Secondary Outcome: Mean Change From Baseline in Disease Activity Score 28 Joints (DAS28) Score
Description: DAS28 is calculated from the number of swollen joints and tender joints using the 28-joints count, the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hr]) and Patient's Global Assessment of Disease Activity (participant-rated arthritis activity assessment) with transformed scores ranging 0 (minimum score) to 10 (maximum score); higher scores indicated greater affectation due to disease activity. A DAS28 score of less than or equal to (=<) 3.2 = low disease activity, a DAS28 score of >3.2 to 5.1 = moderate to high disease activity.
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Rituximab
Number analyzed (Participants) | 72
Units on a scale
  Week 12 (n = 48) | -1.5 (0.2)
  Week 24 (n = 46) | -1.7 (0.2)
Statistical Analysis 1: Comparison: Rituximab; Mean change from Baseline in DAS28 at Week 12: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Rituximab; Mean change from Baseline in DAS28 at Week 24: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p < 0.001, ANOVA

9. Secondary Outcome: Mean Change From Baseline in Patient Global Assessment (100 mm VAS)
Description: The Physician's Global Assessment of disease activity was assessed using a 0 to 100 mm horizontal visual analogue scale (VAS). The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm, as "maximum disease activity" (maximum arthritis disease activity).Change from Baseline = scores at observation minus score at Baseline. An increase in score from Baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Rituximab
Number analyzed (Participants) | 72
Units on a scale
  Week 12 (n = 58) | -25.6 (3.2)
  Week 24 (n = 56) | -23.6 (3.3)
Statistical Analysis 1: Comparison: Rituximab; Mean change from Baseline in patient global assessment at Week 12: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Rituximab; Mean change from Baseline in patient global assessment at Week 24: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p < 0.001, ANOVA

10. Secondary Outcome: Change in HAQ Score From Screening to Weeks 12 and 24
Description: The Health Assessment Questionnaire-Disability Index (HAQ-DI) is a 20-question instrument that assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping and activities of daily living). Responses in each functional area are scored from 0 to 3 (0=no difficulty and 3=inability to perform a task in that area). HAQ-DI total scores expressed as overall mean score with range 0-3: 0-0.25=normal functioning; 0.25-0.5=mild functional limitation; 0.5-1=moderate functional limitation; more than 1=significant functional limitation. The number of participants achieving a clinically important reduction of >= 0.22 point in HAQ (disease-specific questionnaire) at Week 24 was evaluated. HAQ was assessed using the set of observed cases (OC) at each assessment time. An improvement of 0.22 units in HAQ-DI was considered to be a clinically significant improvement.
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Rituximab
Number analyzed (Participants) | 72
Units on a scale
  Week 12 (n = 40) | -0.22 (0.08)
  Week 24 (n = 38) | -0.31 (0.09)
Statistical Analysis 1: Comparison: Rituximab; Change in HAQ score from screening to Week 12: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p = 0.011, ANOVA
Statistical Analysis 2: Comparison: Rituximab; Change in HAQ score from screening to Week 24: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p = 0.001, ANOVA

11. Secondary Outcome: Change in Pain Scale (100-mm VAS) From Screening to Weeks 12 and 24
Description: Visual Analogue Scale (VAS) is a 100 millimeter (mm) scale. Intensity of pain range: 0 mm=no pain to 100 mm=worst possible pain. Change from Screening=scores at observation minus score at Screening. An increase in score from Screening represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement. The change in pain scale was analyzed for the set of observed cases (OC) at each assessment time.
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Rituximab
Number analyzed (Participants) | 72
Units on a scale
  Week 12 (n = 40) | -17.9 (3.7)
  Week 24 (n = 37) | -20.7 (3.6)
Statistical Analysis 1: Comparison: Rituximab; Change in pain scale from screening to Week 12: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Rituximab; Change in pain scale from screening to Week 24: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p < 0.001, ANOVA

12. Secondary Outcome: Change in SF-36 Physical and Mental Component Scores From Screening to Week 12
Description: as for outcome 2
Time Frame: Baseline, Week 12
Population: The ITT population included all screened participants who answered at least one SF-36 questionnaire. n = the number of participants analyzed for a particular component of SF-36.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Rituximab
Number analyzed (Participants) | 72
scores on a scale
  SF-36 Physical component score (n = 39) | 11.2 (3.1)
  SF-36 Mental component score (n = 39) | 10.9 (3.1)
Statistical Analysis 1: Comparison: Rituximab; Physical component score at Week 12: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p = 0.001, ANOVA
Statistical Analysis 2: Comparison: Rituximab; Mental component score at Week 12: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p = 0.001, ANOVA

13. Secondary Outcome: Change in SF-36 Domain Scores From Screening to Week (Wk) 12 and 24
Description: as for outcome 2
Time Frame: Baseline, Week 12, Week 24
Population: The ITT population included all screened participants who answered at least one SF-36 questionnaire. n = the number of participants analyzed for a particular domain of SF-36.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Rituximab
Number analyzed (Participants) | 72
scores on a scale
  Wk 12, Physical functioning domain, n = 39 | 7.2 (4.3)
  Wk 24, Physical functioning domain, n = 38 | 7.6 (2.7)
  Wk 12, Role physical domain, n = 39 | 15.4 (5.5)
  Wk 24, Role physical domain, n = 38 | 21.6 (4.7)
  Wk 12, Bodily pain domain, n = 40 | 14.2 (4.1)
  Wk 24, Bodily pain domain, n = 37 | 17.6 (3.2)
  Wk 12, General health domain, n = 40 | 6.7 (3.7)
  Wk 24, General health domain, n = 37 | 7.7 (4.1)
  Wk 12, Vitality domain, n = 40 | 6.9 (2.8)
  Wk 24, Vitality domain, n = 38 | 7.4 (3.7)
  Wk 12, Social functioning domain, n = 40 | 15 (4.4)
  Wk 24, Social functioning domain, n = 38 | 15.5 (4.9)
  Wk 12, Role emotional domain, n = 39 | 12.4 (4.8)
  Wk 24, Role emotional domain, n = 38 | 7.7 (5.3)
  Wk 12, Mental health domain, n = 40 | 8 (3.4)
  Wk 24, Mental health domain, n = 38 | 8.8 (3.9)
Statistical Analysis 1: Comparison: Rituximab; Physical functioning domain at Week 12: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p = 0.102, ANOVA
Statistical Analysis 2: Comparison: Rituximab; Physical functioning domain at Week 24: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p = 0.008, ANOVA
Statistical Analysis 3: Comparison: Rituximab; Role physical domain at Week 12: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p = 0.008, ANOVA
Statistical Analysis 4: Comparison: Rituximab; Role physical domain at Week 24: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 5: Comparison: Rituximab; Bodily pain domain at Week 12: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p = 0.002, ANOVA
Statistical Analysis 6: Comparison: Rituximab; Bodily pain domain at Week 24: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 7: Comparison: Rituximab; General health domain at Week 12: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p = 0.077, ANOVA
Statistical Analysis 8: Comparison: Rituximab; General health domain at Week 24: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p = 0.068, ANOVA
Statistical Analysis 9: Comparison: Rituximab; Vitality domain at Week 12: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p = 0.018, ANOVA
Statistical Analysis 10: Comparison: Rituximab; Vitality domain at Week 24: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p = 0.053, ANOVA
Statistical Analysis 11: Comparison: Rituximab; Social functioning domain at Week 12: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p = 0.002, ANOVA
Statistical Analysis 12: Comparison: Rituximab; Social functioning domain at Week 24: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p = 0.003, ANOVA
Statistical Analysis 13: Comparison: Rituximab; Role emotional domain at Week 12: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p = 0.015, ANOVA
Statistical Analysis 14: Comparison: Rituximab; Role emotional domain at Week 24: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p = 0.154, ANOVA
Statistical Analysis 15: Comparison: Rituximab; Mental health domain at Week 12: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p = 0.024, ANOVA
Statistical Analysis 16: Comparison: Rituximab; Mental health domain at Week 24: The statistical hypothesis (H0) that the change is equal to 0 is evaluated using the Repeated Measures Analysis of Variance (ANOVA); Test type: Superiority or Other; p = 0.029, ANOVA

14. Secondary Outcome: Percentage of Participants Achieving a Clinically Important Reduction of >= 0.22 Point in HAQ Score at Week 12.
Description: as for outcome 1
Time Frame: Week 12
Population: The ITT population included all screened participants who answered at least one SF-36 questionnaire.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Rituximab
Number analyzed (Participants) | 40
Percentage | 47.5 [32.9 to 62.5]

15. Secondary Outcome: Percentage of Participants Achieving a Clinically Important Increase of >=5 Points in the SF-36 Physical and Mental Component Scores at Weeks 12 and 24.
Description: as for outcome 2
Time Frame: Week 12 and 24
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Rituximab
Number analyzed (Participants) | 72
Percentage
  Physical component score, Week 12, n = 39 | 74.4 [58.9 to 85.4]
  Physical component score, Week 24, n = 36 | 69.4 [53.1 to 82.0]
  Mental component score, Week 12, n = 39 | 74.4 [58.9 to 85.4]
  Mental component score, Week 24, n = 38 | 65.8 [49.9 to 78.8]

ADVERSE EVENTS:
Time Frame: Up to Week 24
Description: An AE was defined as any sign or symptom, including intercurrent illness, that occurred during the course of the study after treatment had started, ie, events that were not present when the participant entered the study or events present at baseline that became worse, whether considered related to treatment or not.
Arm/Group | Rituximab
Serious Adverse Events (participants affected / at risk) | 2/72
Other Adverse Events (participants affected / at risk) | 21/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=72)
Urinary tract infection (Infections and infestations) | 1
Cerebrovascular accident (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=72)
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Influenza (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Secondary syphilis (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Dyspepsia (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
White blood cell disorder (Blood and lymphatic system disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Blood cholesterol increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 2
Phlebitis (Vascular disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.